CLINICAL TRIAL: NCT00447421
Title: Phase I/II Study of Concurrent Cisplatin, Pemetrexed, and Radiotherapy for Limited Stage Small Cell Lung Cancer
Brief Title: A Study to Treat Small Cell Lung Cancer With a Combination of Cisplatin, Pemetrexed, and Radiotherapy
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Interim results of another trial showed inferior activity of treatment
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11089; H3E-EW-S107
Record Dates: First submitted 2007-03-12; First posted 2007-03-14 (Estimated); Results first posted 2009-08-26 (Estimated); Last update posted 2009-10-28 (Estimated); Status verified 2009-10

CONDITIONS: Small Cell Lung Cancer; Carcinoma, Small Cell; SCLC
MeSH Terms: conditions — Small Cell Lung Carcinoma; Carcinoma, Small Cell | interventions — Pemetrexed; Cisplatin; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Drug: pemetrexed; Drug: cisplatin; Radiation: radiation

INTERVENTIONS:
Drug: pemetrexed — Phase 1: 500 mg/m2 then 400 mg/m2, intravenous (IV), every 21 days x 4 cycles (dose escalation)
  Phase 2: 500 mg/m2 then phase 1 determined dose, IV, every 21 days x 4 cycles
  Other Names: LY231514; Alimta
Drug: cisplatin — Phase 1 and Phase 2: 75 mg/m2, intravenous (IV), every 21 days x 4 cycles
Radiation: radiation — Phase 1 and Phase 2: 50-62 Gy, 25-31 days, cycles 2-4

SUMMARY:
The purpose of this study is to determine the recommended dose of pemetrexed, cisplatin and radiotherapy in the treatment of patients with Small Cell Lung Cancer.

ELIGIBILITY:
Inclusion Criteria:

* Measurable disease with diagnosis of Small Cell Lung Cancer.
* Performance status of 0 to 1 on the Eastern Cooperative Oncology Group performance status schedule.
* Patients must be at least 18 years of age and have at least a 12-week life expectancy.
* No prior chemotherapy and/or prior thoracic radiotherapy.
* Adequate pulmonary function and organ function.

Exclusion Criteria:

* Patients with myocardial infarction within the preceding six months.
* Diagnosis of a serious concomitant systemic disorder.
* Prior radiotherapy to the lower neck or abdominal region.
* Significant weight loss.
* Concurrent administration of any other antitumor therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2007-02; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY(1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (4):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leuven, Belgium
- Netherlands (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., 's-Hertogenbosch
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Amsterdam
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rotterdam

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a Phase 1/2 trial that was terminated during Phase 1 and never progressed to Phase 2. The number of patients enrolled is for the Phase 1 portion.
Groups:
- Pemetrexed + Cisplatin: Phase 1: pemetrexed - 500 mg/m2 then 400 mg/m2, intravenous (IV), every 21 days x 4 cycles (dose escalation)
  Phase 2: pemetrexed - 500 mg/m2 then phase 1 determined dose, IV, every 21 days x 4 cycles
  Cisplatin: Phase 1 and Phase 2: 75 mg/m2, intravenous (IV), every 21 days x 4 cycles
  Radiation: Phase 1 and Phase 2: 50-62 gray (Gy), 25-31 days, cycles 2-4
Period: Overall Study
Arm/Group | Pemetrexed + Cisplatin
Started | 9
Completed | 3
Not Completed | 6
Not completed — Lack of Efficacy | 1
Not completed — Adverse Event | 3
Not completed — Sponsor Decision | 2

BASELINE CHARACTERISTICS:
Arm/Group | Pemetrexed + Cisplatin
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 6
Region of Enrollment [Number; unit: participants]
  Belgium | 2
  Netherlands | 7

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Maximum Tolerated Dose
Time Frame: every cycle
Population: This trial was terminated during the Phase 1 portion of this Phase 1/2 trial and it was too early to assess the recommended dose for Phase 2, or to estimate the maximum tolerated dose (MTD).
Measure: Mean (Standard Deviation); unit: milligrams per square meter
Arm/Group | Pemetrexed + Cisplatin
Number analyzed (Participants) | 0

2. Primary Outcome: Phase 2: Overall Response Rate
Description: Overall Response Rate (ORR) was defined as the proportion of participants having either a Complete or Partial response using Response Evaluation Criteria In Solid Tumors (RECIST) criteria. Complete Response=disappearance of all target lesions; Partial Response=30% decrease in sum of longest diameter of target lesions.
Time Frame: baseline to measured progressive disease
Population: This trial was terminated during the Phase 1 portion of this Phase 1/2 trial. No patients were entered into the Phase 2 portion.
Measure: Number; unit: participants
Arm/Group | Pemetrexed + Cisplatin
Number analyzed (Participants) | 0

3. Secondary Outcome: Phase 1: Best Overall Response
Description: Response using Response Evaluation Criteria In Solid Tumors (RECIST) criteria. Complete Response=disappearance of all target lesions; Partial Response=30% decrease in sum of longest diameter of target lesions; Progressive Disease=20% increase in sum of longest diameter of target lesions; Stable Disease=small changes that do not meet above criteria.
Time Frame: baseline to measured response
Population: This trial was terminated during the Phase 1 portion of this Phase 1/2 trial and was stopped too early to assess best overall response.
Measure: Number; unit: participants
Arm/Group | Pemetrexed + Cisplatin
Number analyzed (Participants) | 0

4. Secondary Outcome: Phase 2: Complete Response Rate
Description: Complete Response Rate was defined as the proportion of participants having a Complete Response using Response Evaluation Criteria In Solid Tumors (RECIST) criteria. Complete Response=disappearance of all target lesions.
Time Frame: baseline to measured response time
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Pemetrexed + Cisplatin
Number analyzed (Participants) | 0

5. Secondary Outcome: Phase 2: Time to Progressive Disease
Description: Defined as the time from study enrollment to the first date of disease progression. Time to disease progression was censored at the date of death if death was due to other cause.
Time Frame: baseline to measured progressive disease
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Pemetrexed + Cisplatin
Number analyzed (Participants) | 0

6. Secondary Outcome: Phase 2: Duration of Response
Description: The duration of a complete response (CR) or partial response (PR) was defined as the time from first objective status assessment of CR or PR to the first time of progression or death as a result of any cause.
Time Frame: time of response to progressive disease
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Pemetrexed + Cisplatin
Number analyzed (Participants) | 0

7. Secondary Outcome: Phase 2: Overall Survival
Description: Overall survival was the duration from enrollment to death. For patients who were alive, overall survival was censored at the last contact.
Time Frame: baseline to date of death from any cause
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Pemetrexed + Cisplatin
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Pemetrexed + Cisplatin
Serious Adverse Events (participants affected / at risk) | 6
Other Adverse Events (participants affected / at risk) | 9
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Pemetrexed + Cisplatin
Anaemia (Blood and lymphatic system disorders) | 1/9 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1/9 (1)
Nausea (Gastrointestinal disorders) | 1/9 (1)
Oesophagitis (Gastrointestinal disorders) | 1/9 (1)
Vomiting (Gastrointestinal disorders) | 2/9 (2)
Fatigue (General disorders) | 1/9 (1)
Malaise (General disorders) | 1/9 (2)
Diverticulitis (Infections and infestations) | 1/9 (1)
Lung infection (Infections and infestations) | 1/9 (1)
Pneumonia (Infections and infestations) | 1/9 (1)
Anorexia (Metabolism and nutrition disorders) | 1/9 (1)
Dehydration (Metabolism and nutrition disorders) | 1/9 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1/9 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1/9 (1)
Femoral artery occlusion (Vascular disorders) | 1/9 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk (number of events):
Term (organ system) | Pemetrexed + Cisplatin
Anaemia (Blood and lymphatic system disorders) | 3/9 (3)
Leukopenia (Blood and lymphatic system disorders) | 1/9 (1)
Lymphopenia (Blood and lymphatic system disorders) | 3/9 (3)
Neutropenia (Blood and lymphatic system disorders) | 1/9 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1/9 (1)
Tinnitus (Ear and labyrinth disorders) | 1/9 (1)
Vertigo (Ear and labyrinth disorders) | 1/9 (1)
Lacrimation increased (Eye disorders) | 1/9 (1)
Abdominal pain (Gastrointestinal disorders) | 1/9 (1)
Abdominal pain upper (Gastrointestinal disorders) | 2/9 (2)
Abdominal rigidity (Gastrointestinal disorders) | 1/9 (1)
Constipation (Gastrointestinal disorders) | 3/9 (3)
Diarrhoea (Gastrointestinal disorders) | 4/9 (4)
Dry mouth (Gastrointestinal disorders) | 2/9 (2)
Dyspepsia (Gastrointestinal disorders) | 1/9 (1)
Dysphagia (Gastrointestinal disorders) | 3/9 (3)
Eructation (Gastrointestinal disorders) | 1/9 (1)
Flatulence (Gastrointestinal disorders) | 1/9 (1)
Nausea (Gastrointestinal disorders) | 6/9 (7)
Oesophagitis (Gastrointestinal disorders) | 2/9 (2)
Oral pain (Gastrointestinal disorders) | 1/9 (1)
Stomatitis (Gastrointestinal disorders) | 4/9 (4)
Tongue coated (Gastrointestinal disorders) | 1/9 (1)
Vomiting (Gastrointestinal disorders) | 3/9 (3)
Chest pain (General disorders) | 2/9 (2)
Chills (General disorders) | 1/9 (1)
Fatigue (General disorders) | 4/9 (4)
Injection site reaction (General disorders) | 1/9 (1)
Malaise (General disorders) | 1/9 (1)
Oedema (General disorders) | 1/9 (1)
Oedema peripheral (General disorders) | 1/9 (1)
Pain (General disorders) | 1/9 (1)
Peripheral coldness (General disorders) | 1/9 (1)
Pyrexia (General disorders) | 2/9 (2)
Eye infection (Infections and infestations) | 1/9 (1)
Fungal infection (Infections and infestations) | 1/9 (1)
Lung infection (Infections and infestations) | 1/9 (1)
Nasopharyngitis (Infections and infestations) | 1/9 (1)
Contusion (Injury, poisoning and procedural complications) | 1/9 (1)
Excoriation (Injury, poisoning and procedural complications) | 1/9 (1)
Fall (Injury, poisoning and procedural complications) | 1/9 (1)
Radiation skin injury (Injury, poisoning and procedural complications) | 1/9 (1)
Alanine aminotransferase increased (Investigations) | 1/9 (1)
Creatinine renal clearance decreased (Investigations) | 1/9 (1)
Gamma-glutamyltransferase increased (Investigations) | 1/9 (1)
Glomerular filtration rate decreased (Investigations) | 1/9 (1)
International normalised ratio increased (Investigations) | 1/9 (1)
Neutrophil count decreased (Investigations) | 1/9 (1)
Platelet count decreased (Investigations) | 1/9 (1)
Weight decreased (Investigations) | 1/9 (1)
White blood cell count decreased (Investigations) | 1/9 (1)
Anorexia (Metabolism and nutrition disorders) | 5/9 (5)
Dehydration (Metabolism and nutrition disorders) | 1/9 (1)
Fluid retention (Metabolism and nutrition disorders) | 5/9 (5)
Hyperglycaemia (Metabolism and nutrition disorders) | 1/9 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1/9 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1/9 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 2/9 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 1/9 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 1/9 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1/9 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2/9 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1/9 (1)
Neck mass (Musculoskeletal and connective tissue disorders) | 1/9 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1/9 (1)
Cognitive disorder (Nervous system disorders) | 1/9 (1)
Dizziness (Nervous system disorders) | 2/9 (2)
Dysgeusia (Nervous system disorders) | 2/9 (2)
Headache (Nervous system disorders) | 4/9 (4)
Memory impairment (Nervous system disorders) | 1/9 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1/9 (2)
Anxiety (Psychiatric disorders) | 1/9 (1)
Depressed mood (Psychiatric disorders) | 1/9 (1)
Depression (Psychiatric disorders) | 1/9 (1)
Hallucination (Psychiatric disorders) | 1/9 (1)
Insomnia (Psychiatric disorders) | 3/9 (3)
Restlessness (Psychiatric disorders) | 1/9 (1)
Bladder spasm (Renal and urinary disorders) | 1/9 (1)
Renal failure (Renal and urinary disorders) | 1/9 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1/9 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2/9 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2/9 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1/9 (2)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1/9 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1/9 (1)
Sputum retention (Respiratory, thoracic and mediastinal disorders) | 1/9 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1/9 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1/9 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1/9 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1/9 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 1/9 (1)
Rash (Skin and subcutaneous tissue disorders) | 2/9 (2)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1/9 (1)
Hypotension (Vascular disorders) | 1/9 (1)

LIMITATIONS AND CAVEATS:
The Study Phase 1 was stopped early based on interim results of another trial, showing inferior activity of pemetrexed/carboplatin compared to etoposide/carboplatin in extensive small cell lung cancer. The Study did not progress to Phase 2.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days